CLINICAL TRIAL: NCT06390371
Title: Spotlight AQ Randomized Controlled Trial of the Spotlight AQ Survey Platform to Evaluate Its' Efficacy and Applicability in a Clinic Setting.
Brief Title: Implementing the Spotlight AQ Platform in Adolescent/ Young Adult (16-25 Years Old) Type 1 Diabetics (T1D)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Cintya Schweisberger, Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00002936
Record Dates: First submitted 2024-04-15; First posted 2024-04-30 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Spotlight AQ) (Experimental): Spotlight AQ is an Artificial Intelligence (AI) powered adaptive survey which identifies the main concerns and gaps in patients tailored to their specific needs in preparation for clinic visits
  Interventions: Other: Spotlight AQ Survey platform
- Standard of Care (No Intervention): The pre-clinic survey typically given to patients before clinic visits at each institution

INTERVENTIONS:
Other: Spotlight AQ Survey platform — A psychosocial assessment pinpointing the needs of patients divided into four domains: Therapy, Psychological, Social, Knowledge which is delivered to health care providers to guide their in clinic visits
  Arms: Intervention (Spotlight AQ)

SUMMARY:
The goal of this clinical trial is to compare the Spotlight AQ survey platform to the standard of care (SOC) pre-clinic assessment in adolescents & young adults (16-25 years old) with Type 1 Diabetes (T1D).

The main questions it aims to answer are:

* Does using the Spotlight AQ survey in clinic decrease the A1c in the people who use it?
* Do patients and healthcare providers like using the spotlight AQ survey?

Participants will use the Spotlight AQ survey before coming in to two standard of care T1D clinic visits Participants will fill out surveys describing how they feel about using the Spotlight AQ survey. Some participants may be asked to do an interview to talk about how they feel about the Spotlight AQ survey.

ELIGIBILITY:
Inclusion Criteria:

* 16-25 years old
* Patients diagnosed with T1D for at least 6 months
* On any diabetes treatment
* Using a Continuous Glucose Monitor (CGM)
* Willing/ able to use Spotlight AQ tool
* Able to give verbal assent
* Patients & parents/caregiver speak English/ Spanish fluently
* Patients in the Children's Mercy Kansas City Hospital or Boston Children's Hospital network

Exclusion Criteria:

* <16 years old or >25 years old
* Mental illness that could seriously reduce their ability to participate in the study
* Lack of capacity
* In another T1D intervention study

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 3 months (approximately)
  HbA1c levels of pediatric participants as a %

SECONDARY OUTCOMES:
Participant satisfaction | 3 months (approximately)
  Participant satisfaction with the survey as measured by the End of Study questionnaires. Participants indicate being unsatisfied- satisfied or not helped- helped, etc. within the questionnaires
HCP satisfaction with the Spotlight survey | 3 months (approximately)
  Healthcare Provider (HCP) satisfaction with the Spotlight survey as measured by their End of Study questionnaires. HCPs indicate being unsatisfied- satisfied or not helped- helped, etc. within the questionnaires
T1D outcomes | 3 months (approximately)
  T1D outcomes including Time in Range
T1D outcomes | 3 months (approximately)
  T1D outcomes including bolus scores
The effectiveness of the intervention | 3 months (approximately)
  The effectiveness evaluated in qualitative studies
The approval of participants | 3 months (approximately)
  The approval of participants evaluated in qualitative studies

CONTACTS AND LOCATIONS:
Overall Officials: Cintya Schweisberger, DO, Principal Investigator — Children's Mercy
Locations (1):
- Children's Mercy, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foster NC, Beck RW, Miller KM, Clements MA, Rickels MR, DiMeglio LA, Maahs DM, Tamborlane WV, Bergenstal R, Smith E, Olson BA, Garg SK. State of Type 1 Diabetes Management and Outcomes from the T1D Exchange in 2016-2018. Diabetes Technol Ther. 2019 Feb;21(2):66-72. doi: 10.1089/dia.2018.0384. Epub 2019 Jan 18. PMID 30657336
- [Background] Barnard KD, Lloyd CE, Dyson PA, Davies MJ, O'Neil S, Naresh K, Lawton J, Ziegler R, Holt RI. Kaleidoscope model of diabetes care: time for a rethink? Diabet Med. 2014 May;31(5):522-30. doi: 10.1111/dme.12400. PMID 24506524
- [Background] Reith TP. Burnout in United States Healthcare Professionals: A Narrative Review. Cureus. 2018 Dec 4;10(12):e3681. doi: 10.7759/cureus.3681. PMID 30761233
- [Background] Halbesleben JR, Rathert C. Linking physician burnout and patient outcomes: exploring the dyadic relationship between physicians and patients. Health Care Manage Rev. 2008 Jan-Mar;33(1):29-39. doi: 10.1097/01.HMR.0000304493.87898.72. PMID 18091442
- [Background] Barnard-Kelly K. Utilizing eHealth and Telemedicine Technologies to Enhance Access and Quality of Consultations: It's Not What You Say, It's the Way You Say It. Diabetes Technol Ther. 2019 Jun;21(S2):S241-S247. doi: 10.1089/dia.2019.0015. PMID 31169431
- [Background] Barnard-Kelly K, Kelly RC, Chernavvsky D, Lal R, Cohen L, Ali A. Feasibility of Spotlight Consultations Tool in Routine Care: Real-World Evidence. J Diabetes Sci Technol. 2022 Jul;16(4):939-944. doi: 10.1177/1932296821994088. Epub 2021 Mar 12. PMID 33709795
- [Background] International Diabetes Federation Diabetes Atlas 9th Edition, 2019. https://diabetesatlas.org/en/sections/individual-social-and-economic-impact.html last accessed 16th November 2020
- [Background] Patton SR, Clements MA, Fridlington A, Cohoon C, Turpin AL, Delurgio SA. Frequency of mealtime insulin bolus as a proxy measure of adherence for children and youths with type 1 diabetes mellitus. Diabetes Technol Ther. 2013 Feb;15(2):124-8. doi: 10.1089/dia.2012.0229. Epub 2013 Jan 14. PMID 23317372
- [Background] Kelly RC, Phiri P, Price H, Ali A, Stratton I, Austin K, Neave A, Barnard-Kelly K. Protocol paper: multi-Centre randomised controlled trial evaluating a pre-clinic diabetes assessment and mapped care planning intervention amongst adults with type 1, type 2 or pre-diabetes. Trials. 2022 Jun 20;23(1):515. doi: 10.1186/s13063-022-06475-7. PMID 35725626
- [Background] Patton SR, DeLurgio SA, Fridlington A, Cohoon C, Turpin AL, Clements MA. Frequency of mealtime insulin bolus predicts glycated hemoglobin in youths with type 1 diabetes. Diabetes Technol Ther. 2014 Aug;16(8):519-23. doi: 10.1089/dia.2013.0356. Epub 2014 Apr 28. PMID 24773597
- [Background] Clements MA, DeLurgio SA, Williams DD, Habib S, Halpin K, Patton SR. Association of HbA1c to BOLUS Scores Among Youths with Type 1 Diabetes. Diabetes Technol Ther. 2016 Jun;18(6):351-9. doi: 10.1089/dia.2015.0352. PMID 27258122
- [Background] McConville A, Noser AE, Clements MA, Patton SR. Mealtime insulin BOLUS score increases prior to clinic visits in youth with type 1 diabetes. BMJ Open Diabetes Res Care. 2020 Jul;8(1):e001348. doi: 10.1136/bmjdrc-2020-001348. PMID 32665313